CLINICAL TRIAL: NCT00186836
Title: Efficacy of Combined Hepatitis A and Hepatitis B (Twinrix) Vaccine Compared With Hepatitis B Vaccine Alone in Providing Seroprotection Against Hepatitis B in Hemodialysis Patients
Brief Title: Efficacy Study of Combined Hepatitis A and Hepatitis B Vaccine to Protect Against Hepatitis B in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Health Care London (Other)
Organization: St. Joseph's Healthcare Hamilton (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2400
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Hepatitis B
Keywords: Hepatitis A; Hepatitis B; Hemodialysis; Vaccine
MeSH Terms: conditions — Hepatitis B; Hepatitis A | interventions — Engerix-B; twinrix

INTERVENTIONS:
Biological: Engerix-B and Twinrix

SUMMARY:
Does vaccinating hemodialysis patients with Twinrix® (combination vaccine against hepatitis A and hepatitis B) result in a difference in hepatitis B antibody response in comparison to the monovalent hepatitis B vaccine? Hepatitis B infection is an important cause of mortality and morbidity. Current standard vaccination practices have low efficacy levels in patients (eg. hemodialysis patients) who are most susceptible of infection. Efficacy of the two regiments will be studied.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a human pathogen that causes acute and chronic liver infection. Immunosuppression may be associated with more frequent persistent infection and HBV infections in renal dialysis patients can become chronic. The routes of transmission of the virus is well established; direct percutaneous inoculation of virus via exchange of contaminated blood, blood products, body fluids, and hemodialysis. The Center for Diseases Control and Prevention (CDC) recommends immunization in high-risk groups, including hemodialysis patients. Ninety to ninety five percent of healthy, immunocompent adults develop protective anti-hepatitis B surface antibody (anti-HBs) with a primary series of hepatitis B vaccination, but the overall efficacy in renal dialysis patients is much lower. The proportion of hemodialysis patients who develop a seroprotective antibody even with higher doses of vaccination is a median 64% (range: 34-88%).

Reports suggest that combined vaccination of hepatitis B and hepatitis A (Twinrix®: combination vaccine containing inactivated hepatitis A and recombinant hepatitis B) may improve immunogenicity in healthy individuals. In one study, comparing Anti-HBs geometric mean titres (GMT) at month 6 of the series, subjects receiving the combined vaccine showed a statistically significant higher response than those who obtained the monovalent vaccines. Other studies also reflect the same trend at varying points in the vaccination series.

Currently, there are 426 patients in the hemodialysis program at St. Joseph's Healthcare in Hamilton and 324(76%) patients are susceptible to HBV infection.

Our study will determine if the improved immunogenicity observed with combined HAV and HBV vaccine will increase the efficacy of HBV vaccine in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients
* Age greater than or equal to 18
* Able and willing to give informed consent
* Undetectable Anti-HBs Ab level

Exclusion Criteria:

* Presence of hepatitis BsAg, hepatitis BcAb
* Treatment with IVIg (intravenous immune globulin) within the last 6 months
* Hypersensitivity to components of either vaccine
* Contraindication to intramuscular injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-11; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Hepatitis B antibody response at month 7 (Significant antibody response defined as anti-HBs Ab greater than or equal to 10mIU/mL ).

SECONDARY OUTCOMES:
Anti-HBs geometric mean response at 7 months.
Efficacy of Twinrix® in achieving seroprotection against HAV in hemodialysis patients(Significant antibody response defined as at least 20mIU/mL concentration of anti-HAV.)
Frequency of adverse events associated with vaccine administration

CONTACTS AND LOCATIONS:
Overall Officials: Christine H Lee, MD, Principal Investigator — St. Joseph's Healthcare and McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Murdoch DL, Goa K, Figgitt DP. Combined hepatitis A and B vaccines: a review of their immunogenicity and tolerability. Drugs. 2003;63(23):2625-49. doi: 10.2165/00003495-200363230-00008. PMID 14636084
- [Background] Recommendations for preventing transmission of infections among chronic hemodialysis patients. MMWR Recomm Rep. 2001 Apr 27;50(RR-5):1-43. PMID 11349873
- [Background] Knoll A, Hottentrager B, Kainz J, Bretschneider B, Jilg W. Immunogenicity of a combined hepatitis A and B vaccine in healthy young adults. Vaccine. 2000 Apr 3;18(19):2029-32. doi: 10.1016/s0264-410x(99)00524-1. PMID 10706965
- [Background] Leroux-Roels G, Moreau W, Desombere I, Safary A. Safety and immunogenicity of a combined hepatitis A and hepatitis B vaccine in young healthy adults. Scand J Gastroenterol. 1996 Oct;31(10):1027-31. doi: 10.3109/00365529609003124. PMID 8898425
- [Background] Czeschinski PA, Binding N, Witting U. Hepatitis A and hepatitis B vaccinations: immunogenicity of combined vaccine and of simultaneously or separately applied single vaccines. Vaccine. 2000 Jan 6;18(11-12):1074-80. doi: 10.1016/s0264-410x(99)00354-0. PMID 10590328
- [Background] Abraham B, Baine Y, De-Clercq N, Tordeur E, Gerard PP, Manouvriez PL, Parenti DL. Magnitude and quality of antibody response to a combination hepatitis A and hepatitis B vaccine. Antiviral Res. 2002 Jan;53(1):63-73. doi: 10.1016/s0166-3542(01)00194-2. PMID 11684316
- [Background] Ambrosch F, Andre FE, Delem A, D'Hondt E, Jonas S, Kunz C, Safary A, Wiedermann G. Simultaneous vaccination against hepatitis A and B: results of a controlled study. Vaccine. 1992;10 Suppl 1:S142-5. doi: 10.1016/0264-410x(92)90570-a. PMID 1335647
- [Background] Kallinowski B, Knoll A, Lindner E, Sanger R, Stremmel W, Vollmar J, Zieger B, Jilg W. Can monovalent hepatitis A and B vaccines be replaced by a combined hepatitis A/B vaccine during the primary immunization course? Vaccine. 2000 Aug 15;19(1):16-22. doi: 10.1016/s0264-410x(00)00166-3. PMID 10924782
- [Background] Lee MB, Middleton D. Enteric illness in Ontario, Canada, from 1997 to 2001. J Food Prot. 2003 Jun;66(6):953-61. doi: 10.4315/0362-028x-66.6.953. PMID 12800994
- [Derived] Tung J, Carlisle E, Smieja M, Kim PT, Lee CH. A randomized clinical trial of immunization with combined hepatitis A and B versus hepatitis B alone for hepatitis B seroprotection in hemodialysis patients. Am J Kidney Dis. 2010 Oct;56(4):713-9. doi: 10.1053/j.ajkd.2010.04.015. Epub 2010 Jul 13. PMID 20630640